CLINICAL TRIAL: NCT02180243
Title: CAM in Veterans With Gulf War Illnesses
Acronym: GW-CAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Georgetown University (Other); MedStar Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLD-013-13S; CX000801-01A2 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-10

CONDITIONS: Gulf War Veterans' Illness
Keywords: meditation; acupuncture; Gulf War Veterans' Illness; Gulf War health education; iRest yoga
MeSH Terms: interventions — Mindfulness; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: RBANS assessment was blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness meditation/Acupuncture (Experimental): Eligible participants may be randomized to participate in iRest Yoga Nidra/ auricular acupuncture group classes.
  Interventions: Behavioral: Mindfulness meditation/Acupuncture
- Gulf War Health Education (Active Comparator): Eligible participants may be randomized to participate in Gulf War Health Education group classes.
  Interventions: Other: Gulf War Health Education

INTERVENTIONS:
Behavioral: Mindfulness meditation/Acupuncture — Individuals randomized to this group will participate in iRest Yoga Nidra and auricular acupuncture.
  Arms: Mindfulness meditation/Acupuncture
Other: Gulf War Health Education — Participants randomized to this group will take part in a health education group.
  Arms: Gulf War Health Education

SUMMARY:
The purpose of this study is to explore the effectiveness Gulf War Health Education (GWHE) and iRest Yoga Nidra (mindfulness meditation)/auricular (ear) acupuncture for Veterans with Gulf War Veterans' Illnesses (GWVI).

DETAILED DESCRIPTION:
Gulf War Veterans have reported irritable bowel syndrome, chronic fatigue, musculoskeletal pain, sleep difficulties, and neurocognitive dysfunction (for example, concentration, memory, and attention problems). The most effective treatment approach for what appears to a broad spectrum problem found in GWVI may require complementary alternative medicine (CAM) approaches to enhance positive outcomes. Mindfulness meditation and acupuncture are each broad spectrum CAM treatments designed to target multiple biological systems simultaneously, and thus may be well suited for GWVI. Gulf War Health Education group will promote wellness and prevention by utilizing a proactive patient care model.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veteran
* Deployed to the Gulf War between 1990-1991
* Currently suffers from Gulf War Veterans' Illness (i.e. fatigue, pain, cognitive impairment)

Exclusion Criteria:

* Addiction to drugs or alcohol
* Experiences hallucinations or delusions
* Currently manic
* Currently suicidal
* Hearing difficulties that would interfere with group participation
* Current involvement in a meditation or acupuncture group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Reinhard, PsyD, Principal Investigator — Washington DC VA Medical Center, Washington, DC
Locations (1):
- Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breneman CB, Reinhard MJ, Allen N, Belouali A, Chun T, Crock L, Duncan AD, Dutton MA. Gulf War Illness: A Randomized Controlled Trial Combining Mindfulness Meditation and Auricular Acupuncture. Glob Adv Integr Med Health. 2023 May 3;12:27536130231171854. doi: 10.1177/27536130231171854. eCollection 2023 Jan-Dec. PMID 37151571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between May 2016 and September 2019 via flyers, internet postings with a link to the study recruitment webpage, referrals from primary care providers at the Washington, DC VAMC, and targeted outreach mailings to GW Veterans. Telephone or in-person interviews were conducted to determine eligibility.
Pre-assignment Details: Of 187 Veterans who began the consent process, 37 did not meet inclusion criteria and 1 enrolled but did not complete the randomization procedure. Therefore, 149 Veterans were randomized.
Groups:
- Mindfulness Meditation / Acupuncture: Eligible participants may be randomized to participate in iRest Yoga Nidra/ auricular acupuncture group classes.
  Yoga/Acupuncture: Individuals randomized to this group will participate in iRest Yoga Nidra and auricular acupuncture.
Period: Overall Study
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Started | 75 | 74
Completed | 51 | 60
Not Completed | 24 | 14
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Lost to Follow-up | 12 | 2

BASELINE CHARACTERISTICS:
Population: Some Veterans who completed consent did not complete baseline data collection and were withdrawn from the study at this point.
Groups:
- Mindfulness Meditation / Acupuncture: Eligible participants may be randomized to participate in iRest Yoga Nidra/ auricular acupuncture group.
  Mindfulness meditation /Acupuncture: Individuals randomized to this group will receive iRest Yoga Nidra and auricular acupuncture, administered one right after the other.
- Gulf War Health Education: Eligible participants may be randomized to participate in Gulf War Health Education group.
  Gulf War Health Education: Participants randomized to this group will receive a weekly one-hour education session.
- Total: Total of all reporting groups
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education | Total
Number analyzed (Participants) | 74 | 73 | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.46 (7.15) | 55.16 (7.52) | 54.31 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 57 | 62 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 49 | 53 | 102
  White | 17 | 13 | 30
  Other | 8 | 7 | 15
Education [Mean (Standard Deviation); unit: years] | 14.55 (5.13) | 14.42 (4.51) | 14.49 (4.82)
Married [Count of Participants; unit: Participants] | 47 | 44 | 91
Employed [Count of Participants; unit: Participants] | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Veterans RAND 36-item Health Survey - Mental Component Summary Scale
Description: The MCS is comprised of questions about role-emotional, vitality/mental health and social functioning. Scores are standardized using a t-score transformation and normed to a U.S. population (based on a 1990 norm) of a score of 50 and a standard deviation of 10 where higher scores indicate better health outcomes.
Time Frame: 8 weeks
Population: Participants may have begun but not completed questionnaires assigned via mobile tablet resulting in differences in N for a given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 42.26 (8.56) | 41.75 (8.46)
  Endpoint: number analyzed (Participants) | 51 | 60
  Endpoint | 44.48 (8.09) | 40.62 (8.54)

2. Primary Outcome: Veterans RAND 36-Item Health Survey - Physical Component Summary Scale
Description: The PCS provides emphasis on questions about general health, physical functioning and role playing and bodily pain. Scores are standardized using a t-score transformation and normed to a U.S. population (based on a 1990 norm) of a score of 50 and a standard deviation of 10 where higher scores indicate better health outcomes.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 37.02 (8.78) | 37.00 (10.53)
  Endpoint: number analyzed (Participants) | 51 | 60
  Endpoint | 39.41 (8.78) | 35.69 (10.99)

3. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Adult Short Form v1.0 - Pain Interference 8a
Description: An eight-item self-reported pain instrument designed at the National Institutes of Health (NIH) to measure the extent to which pain interferes with involvement in cognitive, emotional, physical, recreational, and social activities. Higher scores represent greater symptom severity. Range from 0 - 32.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 17.90 (8.96) | 17.47 (9.30)
  Endpoint: number analyzed (Participants) | 51 | 59
  Endpoint | 14.55 (8.14) | 17.77 (9.66)

4. Primary Outcome: Patient-Reported Outcomes Measurement Information System Adult Short Form v1.0 - Fatigue 8a
Description: An 8-item NIH instrument consisting of eight items that asks about the experience and impact of fatigue. Higher scores represent greater symptom severity. Range from 0 - 32.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 20.92 (8.26) | 20.74 (7.64)
  Endpoint: number analyzed (Participants) | 51 | 59
  Endpoint | 17.69 (9.13) | 20.58 (8.65)

5. Secondary Outcome: Short-form McGill Pain Questionnaire (SF-MPQ-2)
Description: The SF-MPQ-2 measures continuous pain, intermittent pain, predominantly neuropathic pain, and affective descriptors. Higher scores indicate greater pain. Symptomatic pain on scale from 0 - 45.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 16.88 (8.75) | 17.01 (9.58)
  Endpoint: number analyzed (Participants) | 51 | 60
  Endpoint | 15.80 (9.46) | 19.42 (10.83)

6. Secondary Outcome: Multidimensional Fatigue Symptom Inventory - Short Form (MFSI-SF)
Description: The MFSI is a 30-item measurement tool that assesses the multidimensional nature of fatigue across five domains: general fatigue, physical fatigue, emotional fatigue, mental fatigue, and vigor. The range is from 24 to 96 with a higher score indicating higher levels of fatigue.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 37.40 (22.56) | 37.78 (23.57)
  Endpoint: number analyzed (Participants) | 51 | 60
  Endpoint | 27.69 (23.15) | 38.17 (27.59)

7. Secondary Outcome: Quality of Life in Neurological Disorders (Neuro-QoL)
Description: The items were selected from the 18 item Neuro-QOL Bank v1.0 - Applied Cognition - General Concerns. Scores range from 1 (very often) to 5 (none) for each cognitive symptom. Higher scores indicate better cognitive function. Range from 18 - 90.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mindfulness Meditation / Acupuncture: Eligible participants may be randomized to participate in iRest Yoga Nidra/ auricular acupuncture group.
  Mindfulness meditation / Acupuncture: Individuals randomized to this group will receive iRest Yoga Nidra and auricular acupuncture, administered one right after the other.
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 48.85 (17.41) | 49.11 (17.77)
  Endpoint: number analyzed (Participants) | 51 | 60
  Endpoint | 55.18 (18.39) | 48.65 (18.99)

8. Secondary Outcome: Patient Health Questionnaire-Depression Module (PHQ-9)
Description: The PHQ is a 9-item questionnaire, used to assess symptoms and functional impairment of depression to derive an overall severity score and a tentative depression diagnosis. Each item score ranges from 0-3 with higher scores indicating more severe depressive symptoms. Range from 0 - 27.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 11.64 (6.42) | 12.29 (7.47)
  Endpoint: number analyzed (Participants) | 50 | 59
  Endpoint | 9.76 (6.86) | 13.32 (8.44)

9. Secondary Outcome: Posttraumatic Symptom Checklist - Civilian Version (PCL-C)
Description: The PCL-C is a 17-item self-report checklist of PTSD symptoms based closely on the DSM-IV criteria with a range of 17-85. Higher scores indicate greater symptom expression.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 31.95 (18.86) | 31.63 (22.04)
  Endpoint: number analyzed (Participants) | 50 | 59
  Endpoint | 26.06 (18.84) | 34.71 (22.66)

10. Secondary Outcome: Perceived Stress Scale (PSS)
Description: The PSS is a 10-item scale that measures the degree to which situations in one's life over the past month are appraised as unpredictable, uncontrollable and overwhelming. Scores range from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 18.68 (7.07) | 18.41 (8.44)
  Endpoint: number analyzed (Participants) | 50 | 59
  Endpoint | 17.24 (6.81) | 19.17 (7.30)

11. Secondary Outcome: The Brief Symptom Inventory (BSI)
Description: The Brief Symptom Inventory is a 53-item self-report inventory in which participants rate the extent to which they have been bothered (0 ="not at all" to 4="extremely") in the past week by various symptoms. Each subscale is averaged for all items, whereby a score of 4 would indicate the highest possible score.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation / Acupuncture | Gulf War Health Education
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 1.12 (0.73) | 1.16 (0.86)
  Endpoint: number analyzed (Participants) | 51 | 60
  Endpoint | 0.97 (0.76) | 1.32 (0.99)

ADVERSE EVENTS:
Time Frame: Adverse events would be collected from baseline (0) until 12 month followups (1 year and 8 weeks from group interventions).
Description: Some Veterans completed consent but did not complete their baseline data collection and were withdrawn from the study at that point.
Arm/Group | Mindfulness Meditation/Acupuncture | Gulf War Health Education
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/73
Other Adverse Events (participants affected / at risk) | 0/74 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT02180243/Prot_SAP_000.pdf